CLINICAL TRIAL: NCT04890873
Title: ERX1000 - A Phase I, Double-blind, Placebo-controlled, Single and Multiple Oral Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study in Male and Female Subjects With Obesity
Brief Title: ERX1000 - Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study in Male and Female Subjects With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ERX Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERX1000-C-002
Record Dates: First submitted 2021-05-07; First posted 2021-05-18 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: ERX1000; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ERX1000 (Experimental): ERX1000 powder provided for preparation of a 4 mg/10 mL oral suspension and 8 mg/10 mL oral suspension
  Proposed dose level for Part A: 4 mg and 8 mg
  Proposed dose level for Part B: 4 and 8 mg. The dose administered will not exceed the highest dose administered in Part A.
  Interventions: Drug: ERX1000
- Placebo (Placebo Comparator): Reference product: Magnesium hydroxide carbonate powder prepared in an oral suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ERX1000 — ERX1000 powder provided for preparation of a 4 mg/10 mL oral suspension and 8 mg/10 mL oral suspension
  Arms: ERX1000
Drug: Placebo — A suspension containing magnesium hydroxide carbonate in polysorbate
  Other Names: Magnesium hydroxide carbonate
  Arms: Placebo

SUMMARY:
The primary objective is to assess the safety and tolerability of single and multiple oral doses of ERX1000 in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.
* Adult females and males, of any race, between 18 and 55 years of age, inclusive, at Screening.
* Females of non-childbearing potential, which is defined as permanently sterile (ie, due to hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), or with bilateral tubal ligation or Essure® (hysteroscopic bilateral tubal occlusion) with confirmation of occlusion of the fallopian tubes performed at least 3 months prior to Screening, or postmenopausal (defined as at least 12 months post cessation of menses without an alternative medical cause and follicle-stimulating hormone [FSH] level

  ≥ 40 mIU/mL). Males will agree to use contraception and refrain from sperm donation.
* Body mass index between 30.0 and 39.9 kg/m^2, inclusive, at Screening.
* Glycosylated hemoglobin (HbA1c) level of < 6.5% at Screening (test may be repeated once for confirmation of out-of-range values).
* Vital signs at Screening and Check-in as per the following ranges and stable (measured in a supine position after a minimum of 5 minutes of rest):

  1. Systolic blood pressure ≥ 90 and ≤ 140 mmHg
  2. Diastolic blood pressure ≥ 50 and ≤ 90 mmHg
  3. Pulse rate ≥ 50 and ≤ 100 bpm.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and/or Check-in as assessed by the Investigator (or designee).

Exclusion Criteria:

* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks prior to dose administration on Day 1.
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* Obesity induced by known endocrine or genetic disorders (eg, Cushing syndrome, hypothyroidism, Prader Willi syndrome).
* Any previous surgical treatment or procedures with medical devices (such as insertion of lap band or gastric balloons) for obesity (excluding liposuction if performed > 1 year prior to Check-in).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, which would increase the subject's risk of participation.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, cholecystectomy, and hernia repair > 6 months prior to Screening will be allowed).
* History or evidence of underlying liver disease, including viral (hepatitis B and C) or alcoholic hepatitis, or confirmed diagnosis of nonalcoholic steatohepatitis (NASH); nonalcoholic fatty liver disease with qualifying liver function tests (LFTs) will be allowed.
* Gilbert's Syndrome (congenital non-hemolytic hyperbilirubinemia) or suspicion of Gilbert's Syndrome based on total and direct bilirubin.
* Laboratory results that exceed the following thresholds at Screening AND Check-in (laboratory tests may be repeated once for confirmation of out-of-range values) as specified:

  1. alanine aminotransferase (ALT) > 1.5 × upper limit of normal (ULN)
  2. aspartate aminotransferase (AST) > 1.5 × ULN
  3. gamma glutamyl transferase (GGT), alkaline phosphatase (ALP), total bilirubin, or International Normalized Ratio (INR) > ULN
  4. Hemoglobinopathy, hemolytic anemia, or chronic anemia (hemoglobin concentration < 13.0 g/dL [130 g/L] for males, < 11.0 g/dL [110 g/L] for females) at Screening or any other condition known to interfere with interpretation of HbA1c measurement
  5. Neutrophils < 1.5 × 109/L deemed clinically significant by Investigator upon a confirmatory repeat
  6. Thyroid-stimulating hormone (TSH) level above the normal range, confirmed on repeat.
* History or presence of cardiac arrhythmia (at the discretion of the Investigator) or congenital long QT syndrome.
* A QT interval corrected for heart rate using Fridericia's method (QTcF) > 450 msec for males or > 470 msec for females on Screening ECG. At the discretion of the Investigator, ECG may be repeated twice and an average taken of the 3 readings.
* The subject has creatinine clearance ≤ 80 mL/minute as calculated using the Cockroft-Gault equation. At the discretion of the Investigator, evaluation may be repeated once to confirm.
* History of alcoholism or drug/chemical abuse within 2 years prior to Check in.
* Alcohol consumption of > 14 units per week. One unit of alcohol equals 12 oz (360 mL) of beer, 1½ oz (45 mL) of liquor, or 5 oz (150 mL) of wine.
* Positive urine drug screen at Screening; or positive alcohol breath test result or positive urine drug screen at Check-in.
* Positive hepatitis B surface antigen and/or hepatitis C antibody and/or positive human immunodeficiency virus 1/2 (Appendix 2).
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives prior to dosing, whichever is longer.
* Subjects who are actively dieting, have gained or lost > 5 pounds, or using or intend to use any prescription or nonprescription drugs for weight loss including herbal or other dietary supplements within 3 months prior to Check-in.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to Check-in and throughout the outpatient Follow-up period.
* Use or intend to use any prescription medications/products within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 14 days prior to Check-in and throughout the outpatient Follow-up period, unless deemed acceptable by the Investigator (or designee).
* Consumption of alcohol from 72 hours prior to Check-in.
* Use of tobacco- or nicotine-containing products (including nicotine and non-nicotine e-cigarettes, vaping, etc.) within 3 months prior to Check-in, or positive cotinine at Screening or Check-in.
* Receipt of blood products within 2 months prior to Check-in.
* Donation of blood from 8 weeks prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
* Poor peripheral venous access.
* Have previously completed or withdrawn from this study or any other study investigating ERX1000, and have previously received the investigational product.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Part A (Single Dose Group A9): Incidence and severity of adverse events (AEs) | Day 1 up to end of study (Day 10)
Part A (Single Dose Group A9): Incidence of clinical laboratory abnormalities | Screening (Day -28) up to end of study (Day 10)
Part A (Single Dose Group A9): Incidence of 12-lead electrocardiogram (ECG) abnormalities | Screening (Day -28 to Day -2), Days 1, 3 and 10
Part A (Single Dose Group A9): Incidence of vital sign abnormalities | Screening (Day -28 to Day -2), Check-in (Day -1), Days 1, 3, 4, 5, 6 and 10
Part A (Single Dose Group A9): Incidence of physical examination abnormalities | Check-in (Day -1), Days 6 and 10
Part B (Multiple Dose Group B5): Incidence of 12-lead electrocardiogram (ECG) abnormalities | Screening (Day -28 to Day -3), Check-in (Day -2), Days 1, 4, 7, 10, 19, 25, 28, 30 and 37
Part B (Multiple Dose Group B5): Incidence of vital sign abnormalities | Screening (Day -28 to Day -3), Check-in (Day -2), Days 1, 3, 4, 5, 6, 7, 9, 10, 11, 12, 13, 14, 15, 16, 19, 22, 25, 28, 30 and 37
Part B (Multiple Dose Group B5): Incidence of physical examination abnormalities | Check-in (Day -2), Days 30, 33 and 37
Part B (Multiple Dose Group B6): Incidence of 12-lead electrocardiogram (ECG) abnormalities | Screening (Day -28 to Day -3), Check-in (Day -2), Days 1, 3, 8, 10, 15, 17, 22, 25, 29, 34 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Incidence of vital sign abnormalities | Screening (Day -28 to Day -3), Check-in (Day -2), Days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 25, 27, 29, 34, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Incidence of physical examination abnormalities | Check-in (Day -2), Days 34, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B5 and Multiple Dose Group B6): Incidence and severity of adverse events (AEs) | Day 1 up to end of study (For Group B5, Day 37 and for Group B6, Day 41)
Part B (Multiple Dose Group B5 and Multiple Dose Group B6): Incidence of clinical laboratory abnormalities | Screening (Day -28), Check-in (Day-2), Days 7, 14, 21, 28, 34 and End of Study (Day 41)

SECONDARY OUTCOMES:
Part A (Single Dose Group A9): Plasma pharmacokinetic (PK) outcome endpoint of ERX1000, AUC0-t | Day 1, 8 and 10
Part A (Single Dose Group A9): Plasma PK outcome endpoint of ERX1000, AUC0-∞ | Day 1, 8 and 10
Part A (Single Dose Group A9): Plasma PK outcome endpoint of ERX1000, AUC0-τ | Day 1, 8 and 10
Part A (Single Dose Group A9): Plasma PK outcome endpoint of ERX1000, Cmax | Day 1, 8 and 10
Part A (Single Dose Group A9): Plasma PK outcome endpoint of ERX1000, Ctrough | Day 1, 8 and 10
Part A (Single Dose Group A9): Plasma PK outcome endpoint of ERX1000, Tmax | Day 1, 8 and 10
Part A (Single Dose Group A9): Plasma PK outcome endpoint of ERX1000, time of last measurable concentration (tlast) | Day 1, 8 and 10
Part A (Single Dose Group A9): Plasma PK outcome endpoint of ERX1000, t1/2 | Day 1, 8 and 10
Part A (Single Dose Group A9): Plasma PK outcome endpoint of ERX1000, apparent total plasma clearance (CL/F) | Day 1, 8 and 10
Part A (Single Dose Group A9): Plasma PK outcome endpoint of ERX1000, apparent volume of distribution (Vz/F) | Day 1, 8 and 10
Part A (Single Dose Group A9): Plasma PK outcome endpoint of ERX1000, accumulation ratio (AR). | Day 1, 8 and 10
Part A (Single Dose Group A9): Urine PK outcome endpoint of ERX1000, amount of drug excreted in urine over the sampling period (Aeu) | Day 1
Part A (Single Dose Group A9): Urine PK outcome endpoint of ERX1000, percentage of dose excreted in urine over the sampling interval (%Feu) | Day 1
Part A (Single Dose Group A9): Urine PK outcome endpoint of ERX1000, renal clearance (CLR) | Day 1
Part B (Multiple Dose Group B5): Plasma pharmacokinetic (PK) outcome endpoint of ERX1000, AUC0-t | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Plasma PK outcome endpoint of ERX1000, AUC0-∞ | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Plasma PK outcome endpoint of ERX1000, AUC0-τ | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Plasma PK outcome endpoint of ERX1000, Cmax | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Plasma PK outcome endpoint of ERX1000, Ctrough | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Plasma PK outcome endpoint of ERX1000, Tmax | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Plasma PK outcome endpoint of ERX1000, time of last measurable concentration (tlast) | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Plasma PK outcome endpoint of ERX1000, t1/2 | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Plasma PK outcome endpoint of ERX1000, apparent total plasma clearance (CL/F) | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Plasma PK outcome endpoint of ERX1000, apparent volume of distribution (Vz/F) | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Plasma PK outcome endpoint of ERX1000, accumulation ratio (AR). | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Urine PK outcome endpoint of ERX1000, amount of drug excreted in urine over the sampling period (Aeu) | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Urine PK outcome endpoint of ERX1000, percentage of dose excreted in urine over the sampling interval (%Feu) | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B5): Urine PK outcome endpoint of ERX1000, renal clearance (CLR) | Days 1, 7, 10, 13, 19, 22, 25, 28, 31, 33 and 37
Part B (Multiple Dose Group B6): Plasma pharmacokinetic (PK) outcome endpoint of ERX1000, AUC0-t | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Plasma PK outcome endpoint of ERX1000, AUC0-∞ | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Plasma PK outcome endpoint of ERX1000, AUC0-τ | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Plasma PK outcome endpoint of ERX1000, Cmax | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Plasma PK outcome endpoint of ERX1000, Ctrough | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Plasma PK outcome endpoint of ERX1000, Tmax | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Plasma PK outcome endpoint of ERX1000, time of last measurable concentration (tlast) | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Plasma PK outcome endpoint of ERX1000, t1/2 | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Plasma PK outcome endpoint of ERX1000, apparent total plasma clearance (CL/F) | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Plasma PK outcome endpoint of ERX1000, apparent volume of distribution (Vz/F) | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Plasma PK outcome endpoint of ERX1000, accumulation ratio (AR). | Days 1, 8, 15, 22, 29, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6): Urine PK outcome endpoint of ERX1000, amount of drug excreted in urine over the sampling period (Aeu) | Day 1 and Day 29
Part B (Multiple Dose Group B6): Urine PK outcome endpoint of ERX1000, percentage of dose excreted in urine over the sampling interval (%Feu) | Day 1 and Day 29
Part B (Multiple Dose Group B6): Urine PK outcome endpoint of ERX1000, renal clearance (CLR) | Day 1 and Day 29
Part B (Multiple Dose Group B5): Pharmacodynamic (PD) outcome endpoint of ERX1000, body weight | Screening (Day -28 to Day -3), Days -1, 8, 15, 22, 28, 30, 33 and 37
Part B (Multiple Dose Group B5): PD outcome endpoint of ERX1000, serum leptin | Days -1, 7, 14, 21, 27 and 30
Part B (Multiple Dose Group B5): PD outcome endpoint of ERX1000, serum lipid - High-density lipoprotein cholesterol (HDL) | Days -1, 14 and 27
Part B (Multiple Dose Group B5): PD outcome endpoint of ERX1000, serum lipid - Low-density lipoprotein cholesterol (LDL) | Days -1, 14 and 27
Part B (Multiple Dose Group B5): PD outcome endpoint of ERX1000, serum lipid -Total cholesterol | Days -1, 14 and 27
Part B (Multiple Dose Group B5): PD outcome endpoint of ERX1000, serum lipid - Triglyceride | Days -1, 14 and 27
Part B (Multiple Dose Group B5): PD outcome endpoint of ERX1000, serum insulin | Days 7 and 21
Part B (Multiple Dose Group B5): PD outcome endpoint of ERX1000, assessment derived from oral glucose tolerance test (OGTT) - serum glucose | Days -1, 14 and 27
Part B (Multiple Dose Group B5): PD outcome endpoint of ERX1000, assessment derived from oral glucose tolerance test (OGTT) - serum insulin | Days -1, 14 and 27
Part B (Multiple Dose Group B5): PD outcome endpoint of ERX1000, derived from oral glucose tolerance test (OGTT) - Homeostatic Model Assessment of Insulin Resistance | Days -1, 14 and 27
Part B (Multiple Dose Group B5): PD outcome endpoint of ERX1000, assessments derived from oral glucose tolerance test (OGTT) - Matsuda Index | Days -1, 14 and 27
Part B (Multiple Dose Group B6):Pharmacodynamic (PD) outcome endpoint of ERX1000, body weight | Screening (Day -28 to -3), Days -1, 1, 8, 15, 22, 29, 34, 36, 38 and End of Study (Day 41)
Part B (Multiple Dose Group B6):PD outcome endpoint of ERX1000, serum leptin | Day -1 and Day 31
Part B (Multiple Dose Group B6): PD outcome endpoint of ERX1000, serum lipid - High-density lipoprotein cholesterol (HDL) | Day -1 and Day 31
Part B (Multiple Dose Group B6): PD outcome endpoint of ERX1000, serum lipid - Low-density lipoprotein cholesterol (LDL) | Day -1 and Day 31
Part B (Multiple Dose Group B6): PD outcome endpoint of ERX1000, serum lipid -Total cholesterol | Day -1 and Day 31
Part B (Multiple Dose Group B6): PD outcome endpoint of ERX1000, serum lipid - Triglyceride | Day -1 and Day 31
Part B (Multiple Dose Group B6):PD outcome endpoint of ERX1000, serum insulin | Day -1 and Day 31
Part B (Multiple Dose Group B6):PD outcome endpoint of ERX1000, assessment derived from oral glucose tolerance test (OGTT) - serum glucose | Day -1 and Day 31
Part B (Multiple Dose Group B6):PD outcome endpoint of ERX1000, assessment derived from oral glucose tolerance test (OGTT) - serum insulin | Day -1 and Day 31
Part B (Multiple Dose Group B6):PD outcome endpoint of ERX1000, assessment derived from oral glucose tolerance test (OGTT) - Homeostatic Model Assessment of Insulin Resistance | Day -1 and Day 31
Part B (Multiple Dose Group B6):PD outcome endpoint of ERX1000, assessments derived from oral glucose tolerance test (OGTT) - Matsuda Index | Day -1 and Day 31

CONTACTS AND LOCATIONS:
Overall Officials: Irene Mirkin, MD, Principal Investigator — Labcorp Clinical Research Unit Inc.
Locations (1):
- Labcorp Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No